CLINICAL TRIAL: NCT03603132
Title: Effects of Different Dosing and Feeding Intervals on the Pharmacokinetic Parameters of Herombopag Olamine Tablets
Brief Title: A Study to Evaluate Different Intervals Between Dosing and Feeding on the Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HR-TPO-Ig
Record Dates: First submitted 2018-06-18; First posted 2018-07-27 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hetrombopag Olamine A (Active Comparator): health subjects received 7.5 mg Hetrombopag Olamine while fasting.
  Interventions: Drug: Hetrombopag Olamine
- Hetrombopag Olamine B (Active Comparator): health subjects received a high-fat meal one hour after taking7.5 mg Hetrombopag Olamine
  Interventions: Drug: Hetrombopag Olamine
- Hetrombopag Olamine C (Active Comparator): health subjects received a high-fat meal two hours after taking7.5 mg Hetrombopag Olamine
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine — 7.5mg in each cycle

SUMMARY:
This study use a single-center, randomized, open, three-cycle, self-control trial design. It is planning to enroll 15 healthy adult male subjects. Fifteen subjects will randomize into 3 test groups which corresponding to 3 different dosing sequences. Subjects will be giving a single oral dose in per cycle, and there will have three types of breakfast administration after each treatment. Washing period is 10 days during the cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. The subject's body weight was ≥ 50.0 kg, BMI was between 19 and 26 kg/m2
3. Signed informed consent.

Exclusion Criteria:

1. Any clinically serious disease that has or is currently suffering from circulatory, endocrine, nervous, digestive, respiratory, hematological, immunological, psychiatric, and metabolic abnormalities, or any other disease that can interfere with the test results
2. Having deep vein thrombosis or other thrombotic diseases.
3. Having thrombocytopenia, mitral valve prolapse, obvious heart murmur, or murmur.
4. Extended QT interval during the screening period (calculated in Bazett's method, males >450 msec)
5. Hepatitis B surface antigen, hepatitis C antibody, syphilis antibody, HIV antibody positive.
6. Those who have a history of allergies to drugs , food or test drugs or similar drugs;
7. Those who have undergone surgery within 4 weeks prior to the trial or plan to perform surgery during the study
8. Those who took any drug within 14 days before the test (including Chinese herbal medicine)
9. Any drug that inhibits or induces liver drug metabolism within 30 days before the test
10. Subjects have participated in other clinical trial within the 3 months prior to study entry.
11. One or more non-pharmacological contraceptive measures cannot be used during the trial, or it is planned to have birth within six months.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Adverse events | from baseline up to Day 26

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | pre-dose ,0.5 h、 1 h、 2 h、 4 h、 6 h、 7 h、 8 h、 10 h、 12 h、 24 h、 48 h、 72 h、 96 h、 120 h after giving dose in each group
Area under the plasma concentration versus time curve (AUC) | pre-dose ,0.5 h、 1 h、 2 h、 4 h、 6 h、 7 h、 8 h、 10 h、 12 h、 24 h、 48 h、 72 h、 96 h、 120 h after giving dose in each group

CONTACTS AND LOCATIONS:
Locations (1):
- The third xiangya hospital Hospital,of central south university, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No